CLINICAL TRIAL: NCT06270940
Title: Prospective Study Upon Pulsed Radiofrequency Therapy on Peripheral Nerves Monitoring Pain, Quality of Life, Patient Satisfaction and Efficacy
Brief Title: Pulsed Radiofrequency Therapy on Peripheral Nerves Monitoring Pain, Quality of Life, Patient Satisfaction and Efficacy
Acronym: PURPOSE
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Katrin Stoecklein, Anesthesiologist, Amsterdam UMC, location VUmc
Other Study IDs: 2023.0922
Record Dates: First submitted 2024-02-02; First posted 2024-02-21 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Prolactin-Releasing Hormone; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pulsed Radiofrequency (PRF) Treatment — PRF treatment maintains a temperature below 42°C and does not produce structural tissue damage around the needle. PRF exposure to the Dorsal Root Ganglion (DRG) induces c-Fos gene expression in the dorsal horn, which suggests a cellular response to the electric forces generated within the DRG. PRF has been found to relieve neuropathic pain by inducing long-term depression of synaptic transmission in the spinal cord, leading to a decrease in allodynia and hyperalgesia. It also modulates the inflammatory response in the injured area by decreasing the expression of pro-inflammatory cytokines, such as TNF-α, in the peripheral nerve and spinal cord, which is a major player in the development and maintenance of neuropathic pain. PRF is characterized by a 500 kHz current applied for 2 pulses per second, with each pulse lasting 20 milliseconds.

SUMMARY:
Neuropathic pain is a chronic condition caused by damage to the somatosensory nervous system. The pain associated with neuropathic pain is often severe and debilitating, and can significantly interfere with the quality of life and daily functioning of affected patients. Current pharmacologic treatments, such as antidepressants, antiepileptics, and opioids, can offer only partial relief for 40-60% of patients, and are often accompanied by severe side effects. This has led to increasing interest in non-pharmacologic management options for neuropathic pain. One such promising treatment option is pulsed radiofrequency (PRF) treatment applied to the affected peripheral nerve in conjunction with local anesthetic and/or corticosteroid medication. Several studies, including case reports, retrospective studies, and small randomized controlled trials, have shown that PRF treatment to the affected peripheral nerve can be beneficial and effective for managing chronic peripheral neuropathic pain. Several peripheral neuralgias, such as thoracic postherpetic neuralgia, occipital neuralgia, pudendal neuralgia, meralgia paresthetica, painful shoulder, post-thoracotomy syndrome, and carpal tunnel syndrome, have been successfully treated with PRF. PRF treatment has garnered significant interest among ultrasound-skilled pain physicians because of its superior, safe, and non-destructive percutaneous approach to peripheral nerves, visualized by today's excellent visual ultrasound guidance. Our academic pain center performs approximately more than 1000 ultrasound-guided peripheral nerve blocks per year on a wide range of peripheral nerves. Moderate evidence for treating peripheral nerves with PRF treatment is available; however, PRF treatment settings such as voltage, number of cycles, and treatment duration vary, and it is not clear which setting contributes most substantially to pain reduction results. The aim of this prospective longitudinal observational data collection is to evaluate the efficacy of PRF treatment applied to peripheral nerves, to observe the clinical course of chronic peripheral neuropathic pain under conditions of routine clinical practice, and to link these observations with clinical outcomes.

DETAILED DESCRIPTION:
Patients with chronic peripheral neuropathic pain visiting the outpatient pain clinic and who will be scheduled for PRF treatment will be considered for inclusion by the treating pain physician. When meeting the inclusion criteria and none of the exclusion criteria, the patient will receive verbal information (during the patient visit or by phone) and will be asked to participate in this data collection. Signed informed consent will be obtained during the outpatient pain clinic consultation.

This study follows a Data Management Plan which provides relevant information regarding data management requirements.

A) Study Preparation: The dataset is encoded via a unique, meaningless code (Subject ID). Data are de-identified within the study database. Data acquisition has been registered with the Data Protection Officer (DPO). An informed consent procedure has been established that describes the dataset, the timeframe for data retention, information on data sharing, and making data available for future research. A central location for all digital and hard copy study documents exists.

B) Data acquisition: Reuse of existing data, such as patient characteristics in the patient's medical record system in EPIC, is covered by the subject's informed consent.

C) Data collection: The Castor EDC system is used for data collection. Licensing and processing agreements have been arranged. The researchers are trained in using this system, and documentation of their training is available. The database was designed before being built, and a data dictionary was created. Validation checks for completeness, correctness, and consistency are incorporated into the data collection system and have been documented. The data collection system has been tested by both the study team and an independent party. Access to the data collection system is based on individual login with only the necessary access rights and is managed under supervision and documented by the Principal Investigator (PI). Users are trained in the data collection system.

D) Data storage: Raw, interim, final, and key files are stored on the department's M-drive. Raw and final files are stored on the data storage facility at Amsterdam University Medical Center and on the Castor storage facility.

E) Data collection: A site signature and delegation log of all people involved in the data collection are kept by the PI. Checks for completeness, correctness, and consistency are built into the system. An audit trail and track changes functionality are used in the applied system. All changes in the design will be documented to ensure an impact assessment of these changes is performed. Approval and the reason for locking the data collection have been documented.

F) Processing and statistical analysis: The data are stored in a generic and machine-actionable format, such as CSV, and also stored in SPSS as a read-only file. All data processing and analysis are programmed in syntax or script files.

G) Writing and publishing: For each manuscript, a structured subfolder has been created.

H) Data sharing and archiving: Metadata (documentation on study procedures, data dictionary, data validation, and derivation plan) and final data will be published. For verification purposes, all data are stored internally. A de-identified dataset will be made available upon request to the corresponding author. The request must include ethics approval and a statistical analysis plan. The embargo period is at least 1 year after the publication of the original study. For data reuse, a Data Sharing Agreement will be set up. Digital data (metadata, raw data files, final data files), and documentation will be preserved for 10 years. A subject identification log is archived and kept separate from other study-related data. This does not conflict with the subject's informed consent. Paper documentation will be preserved for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18
* Dutch speaking
* Chronic peripheral neuropathic pain lasting ≥ 6 months with mean NRS pain score of ≥ 4
* Patients who are scheduled for an ultrasound guided PRF treatment on a peripheral nerve
* Willing and able to sign consent

Exclusion Criteria:

- Inability to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this data collection consists of patients who will receive PRF treatment for chronic peripheral neuropathic pain (duration of pain ≥ 6 months).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Duration PRF | Procedure
  Duration PRF: 4 or 8 minutes
Type of PRF | Procedure
  2 Hz of 5 Hz / 5 ms or 20 ms / Monopolar or bipolar / Voltage / Temperature / Resistance / Current
Pain intensity | Baseline, 6 weeks, 3 months, 6 months
  Pain with NRS (Numeric Rating Scale): Min=0 / Max=10 / Low score is better
Health Related Quality of life | Baseline, 6 weeks, 3 months, 6 months
  EQ-5D-5L (EuroQol Quality of life) questionnaire: Index=Patient health state / Min=-0.446 / Max=1 / Higher is better / Patient self rated health: Min=0% / Max=100% / High scores are better
Patient Global Impression of Change: PGIC | 6 weeks, 3 months, 6 months
  Patient Global Impression of Change: 7-point likert scale / Much better to much worse
Use of opioids | Baseline, 6 weeks, 3 months, 6 months
  Change of opioid medication (mg) / Min=0 mg / Max=not set / Lower values are better
PROMIS-29 | Baseline, 6 weeks, 3 months, 6 months
  PROMIS: Profile-29 questionnaire; Standardized t-scoring with mean=50 and SD=10 in Dutch reference population
PROMIS Global-10 | Baseline, 6 weeks, 3 months, 6 months
  ROMIS Global 10: Consists of ten (10) items that measure physical health, physical functioning, general mental health, emotional distress, satisfaction with social activities and relationships, ability to carry out usual social activities and roles, pain, fatigue and overall quality of life. Standardized t-scoring with mean=50 and SD=10 in Dutch reference population.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Steegers, Prof, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No